CLINICAL TRIAL: NCT00800371
Title: Diagnostic Value of MRI and Ultrasound in Patients With JIA
Brief Title: Magnetic Resonance Imaging (MRI) in Asymptomatic Patients With Juvenile Idiopathic Arthritis (JIA)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Nikolay Tzaribachev, MD, University Children's Hospital
Other Study IDs: Silent Arthritis PROSPECT 2008
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-11

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: JIA
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- JIA: Patients with JIA
  Interventions: Procedure: intra-articular steroid injection

INTERVENTIONS:
Procedure: intra-articular steroid injection — Steroid injection into otherwise noncontrollable arthritis.

SUMMARY:
Juvenile idiopathic arthritis (JIA) may progress asymptomatically leading to joint destruction despite treatment.

The aim of the observational study is to describe patients with silent arthritis comparing symptoms, clinical findings with results of ultrasound and magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* children without symptoms or with only mild joints swelling or with only minimal limited range of motion

Exclusion Criteria:

* patients with manifest arthritis

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with JIA
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Definition of patients with silent arthritis. | every three to six months from recruitment to end of study

SECONDARY OUTCOMES:
Comparison of diagnostic value of MRI and ultrasound. | every three to six months from recruitment to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay Tzaribachev, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Children's Hospital, Tübingen, Baden-Wurttemberg, Germany